CLINICAL TRIAL: NCT02847143
Title: A Cross Over Randomized Controlled Trial of the Effect of Nasal Ocytocine on Cerebral Activations in Relation With Attachement in the General Population
Brief Title: Ocytocine and Cerebral Activation in Relation With Attachement
Acronym: OTACLA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P/2014/237
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2021-06

CONDITIONS: Attachement Style
Keywords: Attachement; Oxytocin; fMRI
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- secure (Experimental): healthy adult male with secure attachement
  Interventions: Drug: nasal oxytocin or placebo; Device: fMRI; Behavioral: Attachement scale interview (ASI); Behavioral: psychometric scales
- avoidant (Experimental): healthy adult male with avoidant attachement
  Interventions: Drug: nasal oxytocin or placebo; Device: fMRI; Behavioral: Attachement scale interview (ASI); Behavioral: psychometric scales
- enmeshed/fearfull (Experimental): healthy adult male with enmeshed/fearfull attachement
  Interventions: Drug: nasal oxytocin or placebo; Device: fMRI; Behavioral: Attachement scale interview (ASI); Behavioral: psychometric scales
- dual style (Experimental): healthy adult male with dual attachement style
  Interventions: Drug: nasal oxytocin or placebo; Device: fMRI; Behavioral: Attachement scale interview (ASI); Behavioral: psychometric scales

INTERVENTIONS:
Drug: nasal oxytocin or placebo — nasal administration of oxytocin or palcebo 45 min befor fMRI session
Device: fMRI — FMRI during emotional image visualization
Behavioral: Attachement scale interview (ASI) — this scale is used to determine the attachement style of each participant
Behavioral: psychometric scales — self adminstrated questionnaires which asses the level of anxiety (Spielberger State-trait anxiety interview-STAI), depression (Beck depression inventory-BDI) and alexithymia (Toronta Alexuthymia scale-TAS 20)

SUMMARY:
The study aims to characterize the cerebral activation modifications related to nasal oxytocin administration during vizualisation of distress images in population of healthy people with different attachement styles.

DETAILED DESCRIPTION:
Healthy adult male will be recruited. Their attachement style will be assessed through the Attachement scale interview (ASI).

They will have 2 fMRI sessions, during which emotional images will be presented.

One session will be preceded by a nasal administration of oxytocin and the other session will be preceded by a placebo nasal administration. The order of both administrations will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* comprehension of french
* having signed the informed consent

Exclusion Criteria:

* chronic disease (liver failure, kidney failure) and cardiovascular disease
* hypertensive treatment
* treatment wich increases QT
* current hospitalisation
* fMRI contraindication
* legal protection

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
BOLD signal intensity | 45 min after intranasal administration of oxytocin or placebo
  BOLD signal will be assessed in the brain regions associated with attachement: amygdala, medial prefrontal cortex and dorsolateral prefrontal cortex.
  Both conditions (placebo vs axytocin) will be compared in the four groups. BOLD signal will be assessed during the visualization of emotional pictures that ellicit distress, comfort or complicity or neural emotion.

CONTACTS AND LOCATIONS:
Overall Officials: Lauriane VULLIEZ-COADY, MD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Comte A, Szymanska M, Monnin J, Moulin T, Nezelof S, Magnin E, Jardri R, Vulliez-Coady L. Neural correlates of distress and comfort in individuals with avoidant, anxious and secure attachment style: an fMRI study. Attach Hum Dev. 2024 Oct;26(5):423-445. doi: 10.1080/14616734.2024.2384393. Epub 2024 Aug 2. PMID 39093338